CLINICAL TRIAL: NCT02783508
Title: Pethidine Versus Nitrous Oxide for Pain Relief During Labor Among Multiparous. A Randomized Controlled Trial
Brief Title: Pethidine Versus Nitrous Oxide for Pain Relief During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Sivan Easton, Medical Doctor, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0072-016-EMC
Record Dates: First submitted 2016-05-18; First posted 2016-05-26 (Estimated); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Labor Pain
Keywords: Labor analgesia; Nitrous Oxide; Meperidine; Multiparous; Visual analogue scale
MeSH Terms: conditions — Labor Pain | interventions — Meperidine; Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Meperidine (Active Comparator): Intravenous injection of meperidine 50mg given in 100cc NaCl 0.9% over 10 minutes. Repeated doses (if needed) will be given in intervals of 2 hours minimum until a maximum of 4 doses.
  Interventions: Drug: IV Meperidine
- Inhaled Nitrous Oxide (Active Comparator): Nitrous oxide in a 50/50 mix with oxygen given via self-administered face mask. The parturient will be advised to place the mask tightly on her face and to breathe through it at the first sign of forthcoming uterine contraction. Between contractions, the parturient will be advised not to breath through the mask.
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: IV Meperidine — Intravenous meperidine 50mg in 100cc NaCl 0.9% . Repeated doses (if needed): intervals of 2 hours minimum until a maximum of 4 doses.
  In cases of nausea or vomiting intravenous metoclopramide 10mg will be offered to the parturient.
  If pain intensity (according to visual analogue scale), 20 to 30 minutes from administration, will not decline or the parturient will ask for a different type of analgesia, inhaled nitrous oxide or epidural analgesia will be offered.
  Other Names: Pethidine
  Arms: IV Meperidine
Drug: Nitrous Oxide — Nitrous oxide in a 50/50 mix with oxygen given via self-administered face mask. The parturient will be advised to place the mask tightly on her face and to breathe through it at the first sign of forthcoming uterine contraction. Between contractions, she will be advised not to breathe through the mask.
  In cases of nausea or vomiting intravenous metoclopramide 10mg will be offered to the parturient.
  If pain intensity (according to visual analogue scale), 20 to 30 minutes from administration, will not decline or the parturient will ask for a different type of analgesia, intravenous meperidine or epidural analgesia will be offered.
  Other Names: N2O
  Arms: Inhaled Nitrous Oxide

SUMMARY:
Systematic opioids and inhaled nitrous oxide (N2O ) are common methods for pain relief during labor. The aim of the current study is to evaluate the efficacy of systemic pethidine compared to N2O given for pain relieve in term, multiparous women in labor.

DETAILED DESCRIPTION:
Pain relief during labor and delivery is an essential part of good obstetrical care. Labor pain and its relief have implications on the course of labor, maternal and fetal outcomes and the satisfaction with childbirth overall. Many women would like to have a choice in pain relief during labor but also would like to avoid invasive methods of pain management in labor (as epidural). Both, inhaled analgesia and parenteral opioids are common pharmacological interventions aim to relieve the pain of labor.Nitrous oxide in a 50/50 mix with oxygen is the most common concentration used for labor pain management. It is self-administered via facemask, intermittently, and has rapid onset and offset effect. Main side effects, including nausea, vomiting, dizziness and drowsiness. Pethidine is one of the most frequently used opiate agonists. It can be given intravenous or intramuscularly. Its analgesic effect starts within 10-20 minutes and lasts 2-4 hours. Reported maternal side effects include nausea, vomiting and dysphoria. Pethidine may lead to changes in fetal heart rate tracing during labor, respiratory depression, impaired sucking reflex and restlessness.

Given the fact that these two routine interventions are given in different ways and have different side effects profile, the investigators aim in this randomized controlled trial to compare the analgesic effect of these two methods and their maternal and perinatal secondary effects in multiparous laboring women.

ELIGIBILITY:
Inclusion Criteria:

1. Multiparity (para 2 or more).
2. Term pregnancy: 37-42 weeks of gestation.
3. Singleton pregnancy.
4. Vertex presentation.
5. In labor: at least 2 contraction in ten minutes and cervical dilatation of 2 centimeters or more.

Exclusion Criteria:

1. Women who desire epidural as a first line analgesia during labor.
2. Women receiving pethidine during the last 24 hours (prior to entering labor room).
3. Contra-indication for vaginal delivery.
4. Contra-indication or allergic reaction to either pethidine or nitrous oxide.
5. History of drug abuse.
6. Previous cesarean delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 20-30 minutes after drug administration.
  Visual analogue scale

SECONDARY OUTCOMES:
Pain intensity | 60, 120 and 180 minutes from drug administration.
  Visual analogue scale
Time from drug administration to labor. | 24 hours
Need for additional analgesia | 24 hours
  Number of women that needed additional analgesia.
Side effects. | During 60 minutes from drug administration.
  nausea, vomiting, itching, headache, mouth dryness, drowsiness
Breast feeding | Up to 48 hours after birth
Participants satisfaction and the usefulness of pain relief | Within 48 hours after birth
  Scale of excellent, very good, good, fair or poor.
Changes in electronic fetal heart rate monitoring | 24 hours
Occurence of meconium stained amniotic fluid | 24 hours
  Number of women with meconium stained amniotic fluid.
Umbilical artery PH | Up to 5 min from birth, after performing cord clamping.
  Number of women with Umbilical artery PH less than 7.1.
Apgar score | At 1 and 5 minutes after birth
Need for respiration | Within 48 hours after birth
Neonatal Intensive Care Unit (NICU) administration | Within 48 hours after birth
  Number of neonates that admitted to neonatal intensive care unit within 48 hours after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — haemek medical center; Sivan Easton, MD, Principal Investigator — haemek medical center
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klomp T, van Poppel M, Jones L, Lazet J, Di Nisio M, Lagro-Janssen AL. Inhaled analgesia for pain management in labour. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD009351. doi: 10.1002/14651858.CD009351.pub2. PMID 22972140
- [Background] Keskin HL, Keskin EA, Avsar AF, Tabuk M, Caglar GS. Pethidine versus tramadol for pain relief during labor. Int J Gynaecol Obstet. 2003 Jul;82(1):11-6. doi: 10.1016/s0020-7292(03)00047-x. PMID 12834936
- [Background] Likis FE, Andrews JC, Collins MR, Lewis RM, Seroogy JJ, Starr SA, Walden RR, McPheeters ML. Nitrous oxide for the management of labor pain: a systematic review. Anesth Analg. 2014 Jan;118(1):153-67. doi: 10.1213/ANE.0b013e3182a7f73c. PMID 24356165
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Wee MY, Tuckey JP, Thomas PW, Burnard S. A comparison of intramuscular diamorphine and intramuscular pethidine for labour analgesia: a two-centre randomised blinded controlled trial. BJOG. 2014 Mar;121(4):447-56. doi: 10.1111/1471-0528.12532. Epub 2013 Dec 2. PMID 24289216
- [Background] Howell CJ, Kidd C, Roberts W, Upton P, Lucking L, Jones PW, Johanson RB. A randomised controlled trial of epidural compared with non-epidural analgesia in labour. BJOG. 2001 Jan;108(1):27-33. doi: 10.1111/j.1471-0528.2001.00012.x. PMID 11213000
- [Background] Macones GA, Hankins GD, Spong CY, Hauth J, Moore T. The 2008 National Institute of Child Health and Human Development workshop report on electronic fetal monitoring: update on definitions, interpretation, and research guidelines. Obstet Gynecol. 2008 Sep;112(3):661-6. doi: 10.1097/AOG.0b013e3181841395. PMID 18757666
- [Derived] Zuarez-Easton S, Zafran N, Garmi G, Dagilayske D, Inbar S, Salim R. Meperidine Compared With Nitrous Oxide for Intrapartum Pain Relief in Multiparous Patients: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jan 1;141(1):4-10. doi: 10.1097/AOG.0000000000005011. Epub 2022 Dec 2. PMID 36701604